CLINICAL TRIAL: NCT01103193
Title: Nitrous Oxide - Sevoflurane-Remifentanil Interaction: Multiple Response Surfaces, Validation of Calibration Stimuli, Validation of the Intraoperative Isobole Concept and Investigating Remifentanil Induced Opioid Tolerance.
Brief Title: Nitrous Oxide - Sevoflurane-Remifentanil Interaction
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Need of change to the protocol. As the Principal Investigator has left the University Hospital Ghent end 2010, the change of protocol was never submitted.
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009/493
Record Dates: First submitted 2010-03-19; First posted 2010-04-14 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2012-05

CONDITIONS: ASA Class I/II Patients Scheduled for Surgery Under General Anesthesia
Keywords: ASA class I/II patients, with surgery under general anesthesia
MeSH Terms: interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- remifentanil injected (Active Comparator): a mixture of 60% nitrous oxide and 40% oxygen is administered through a face mask. In the first group the patient receives a constant concentration of sevoflurane. In this group the remifentanil concentration will be injected via an intravenous line in a step up protocol.
  Interventions: Drug: remifentanil injected
- sevoflurane in step up concentration (Active Comparator): a mixture of 60% nitrous oxide and 40% oxygen is administered through a face mask. remifentanil is injected in a fixed rate and sevoflurane is administered in a step up concentration.
  Interventions: Drug: sevoflurane in step up concentration

INTERVENTIONS:
Drug: remifentanil injected — mixture of 60% nitrous oxide and 40% oxygen is administered through a face mask. In the first group the patient receives a constant concentration of sevoflurane. In this group the remifentanil concentration will be injected via an intravenous line in a step up protocol.
  Arms: remifentanil injected
Drug: sevoflurane in step up concentration — of 60% nitrous oxide and 40% oxygen is administered through a face mask.remifentanil is injected in a fixed rate and sevoflurane is administered in a step up concentration.
  Arms: sevoflurane in step up concentration

SUMMARY:
patients are allocated to one of the two study groups.

In both groups a mixture of 60% nitrous oxide and 40% oxygen is administered through a face mask. In the first group the patient receives a constant concentration of sevoflurane. In this group the remifentanil concentration will be injected via an intravenous line in a step up protocol. In the second group remifentanil is injected in a fixed rate and sevoflurane is administered in a step up concentration.

During the study, at predefined times, we will assess different levels of sedation (OAA/S score) and the reaction on tetanic stimulation of the ulnar nerve, insertion of a laryngeal mask airway and laryngoscopy. In addition heart rate, SpO2 and capnography will be recorded continuously and non invasive bloodpressure will be recorded using a 1 minute interval time. Spectral entropy and BIS derived from the frontal EEG will be used to monitor clinical cerebral drug effect.

The null hypothesis is that remifentanil lowers the concentration of sevoflurane dissolved in a mixture of 60% nitrous oxide and 40% oxygen to (1) tolerate a specific stimulation and to (2) obtain a certain electroencephalographic parameter value and vice versa. Additionally the results of this study will be compared with a former interaction study of the same study group that did not involve nitrous oxide, in order to depict the shift in the response surface evoked by nitrous oxide.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesia class I and II patients
* aged 18-60 years
* scheduled for surgery under general anesthesia.

Exclusion Criteria:

* Weight less than 70% or more than 130% of ideal body weight
* neurological disorder
* diseases involving the cardiovascular system, pulmonary disease, gastric diseases, endocrinological diseases
* recent use of psycho-active medication, including alcohol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2010-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To investigate the pharmacodynamic interaction between nitrous oxide, sevoflurane and remifentanil | Every 12 minutes during induction and maintenance of anesthesia
  The interaction is studied on response surfaces including several clinical endpoints: the observer assessment of alertness and sedation scale, the heart rate, pulse oximetry, blood pressure, EEG and the derived parameters from it: spectral entropy and BIS

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Vereecke, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: website University Hospital Ghent — http://www.uzgent.be